CLINICAL TRIAL: NCT07159165
Title: Minimal Invasive Urology Society Benign Prostatic Obstruction (BPO) Study Group Data Collection Project
Brief Title: Registry of MIUS for Benign Prostatic Obstruction
Acronym: ReMIUS-BPO
Status: Enrolling by invitation | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Ankara University (Other); Dokuz Eylul University (Other); Erol Olcok Corum Training and Research Hospital (Other); Gazi University (Other); Eskisehir Osmangazi University (Other); Marmara University (Other); Samsun Education and Research Hospital (Other); Cukurova University (Other); Izmir Metropolitan Municipality Esrefpasa Hospital (Unknown); Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Murat Gulsen, Assistant Professor, Ondokuz Mayıs University
Other Study IDs: MIUS.2025.001
Record Dates: First submitted 2025-08-08; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia With Lower Urinary Tract Symptoms
Keywords: Benign Prostatic Obstruction; Lower Urinary Tract Symptoms; Prostatic Surgery; Transurethral Resection of the Prostate; Holmium Laser Enucleation of the Prostate; Thulium Laser Enucleation of the Prostate; Rezum; Minimally Invasive Surgery; Laser Enucleation; Prostate Endoscopic Surgery; Urology; Prospective Registry; Multicenter Study; BPO; LUTS; TURP; HoLEP; ThuLEP
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing minimally invasive surgical treatment for BPO: All eligible male patients with a diagnosis of BPO undergoing procedures such as TURP, HoLEP, ThuLEP, Rezum®, or similar minimally invasive techniques will be included.
  Interventions: Procedure: Minimally invasive surgical treatment for benign prostatic obstruction

INTERVENTIONS:
Procedure: Minimally invasive surgical treatment for benign prostatic obstruction — Surgical management of BPO using contemporary minimally invasive procedures, including but not limited to: Transurethral resection of the prostate (TURP), Holmium laser enucleation of the prostate (HoLEP), Thulium laser enucleation of the prostate (ThuLEP), Rezum® water vapor thermal therapy.
  Procedures are performed according to standard clinical practice at each participating center, with perioperative and follow-up data prospectively recorded in the MIUS registry.

SUMMARY:
This national, multicenter, prospective registry aims to collect standardized perioperative and follow-up data on patients undergoing minimally invasive surgical management for benign prostatic obstruction (BPO) in Turkey. Procedures include transurethral resection of the prostate (TURP), holmium/thulium laser enucleation (HoLEP/ThuLEP), Rezum®, and other contemporary techniques. By prospectively recording patient characteristics, surgical details, and postoperative outcomes in a unified electronic database, the project seeks to provide high-quality real-world evidence to support clinical decision-making, guideline updates, and future hypothesis-driven sub-studies.

DETAILED DESCRIPTION:
The ReMIUS-BPO registry is designed as a prospective, observational, multicenter cohort study under the coordination of the Minimal Invasive Urology Society. Participating centers will record preoperative, intraoperative, and postoperative data of patients undergoing minimally invasive surgery for BPO using a secure, standardized electronic case report form. Preoperative variables include demographics, comorbidities, medication history, prostate volume, and validated symptom scores (IPSS, OAB-V8). Intraoperative data include surgical technique, energy source, operative time, and complications. Postoperative follow-up will record early and late complications, catheterization time, changes in symptom scores, and re-intervention rates.

The registry aims to:

1. Create a comprehensive, analyzable national dataset for BPO surgery.
2. Compare surgical outcomes between different energy sources.
3. Evaluate the impact of the learning curve on operative time.
4. Determine long-term reoperation rates. The data will serve as a platform for future hypothesis-driven studies and potential embedded randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Male patients ≥ 18 years old
* Diagnosis of BPO with clinical indication for minimally invasive surgery
* Signed informed consent
* Availability of complete baseline and follow-up data

Exclusion Criteria:

* No informed consent
* Missing essential preoperative or follow-up data

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult male patients (≥18 years) diagnosed with benign prostatic obstruction (BPO) and scheduled to undergo minimally invasive surgical treatment at participating centers. The registry will include consecutive eligible patients treated with procedures such as transurethral resection of the prostate (TURP), holmium laser enucleation of the prostate (HoLEP), thulium laser enucleation of the prostate (ThuLEP), Rezum®, or other contemporary surgical techniques, according to routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible BPO surgery patients successfully enrolled with complete baseline, perioperative, and follow-up data in the MIUS registry | Within 12 months after each patient's surgery date
  Percentage of eligible patients undergoing minimally invasive surgical treatment for BPO whose data sets are complete for all predefined variables (baseline characteristics, perioperative details, and follow-up outcomes) in the national MIUS registry. Completeness is defined as ≥95% of required data fields filled for each case.

SECONDARY OUTCOMES:
Comparison of perioperative complication rates between surgical techniques | up to 4 weeks
  Proportion of patients experiencing perioperative complications (Clavien-Dindo classification) following TURP, HoLEP, ThuLEP, or Rezum®
Change in International Prostate Symptom Score (IPSS) | Baseline to 12 months post-surgery
  Mean change in International Prostate Symptom Score (IPSS) from baseline to 12 months in patients undergoing minimally invasive surgical treatment for benign prostatic obstruction (BPO).
  The IPSS ranges from 0 to 35, with higher scores indicating more severe lower urinary tract symptoms (worse outcome).
Change in maximum urinary flow rate (Qmax) | Baseline to 12 months post-surgery
  Mean difference in Qmax (mL/sec) between preoperative measurement and 12-month follow-up.
Reoperation-free survival | Up to 5 years post-surgery
  Proportion of patients not requiring repeat surgical intervention for BPO within 5 years after the index procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and data protection regulations, including the Turkish Personal Data Protection Law (KVKK). Only aggregated, de-identified results will be reported in publications and presentations.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT07159165/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT07159165/ICF_001.pdf